CLINICAL TRIAL: NCT02050802
Title: A Double-blind, Randomized, Placebo-controlled, Four-way Crossover Phase 1 Study Including an Open-label Positive Control (Moxifloxacin) to Assess the Effect of Repeated Daily Doses of 10 mg and 30 mg Macitentan on the QT/QTc Interval of the ECG in Healthy Male and Female Subjects
Brief Title: Study to Assess the Effect of Macitentan on the Electrocardiogram (ECG) in Healthy Male and Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: AC-055-114
Record Dates: First submitted 2014-01-29; First posted 2014-01-31 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy
Keywords: Macitentan; Pharmacokinetics; Pharmacodynamics
MeSH Terms: interventions — Moxifloxacin; macitentan

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (8):
- Treatment sequence BCAD (Experimental): Subjects received study medication in the sequence BCAD. Treatment A: moxifloxacin positive control (3 placebo tablets once daily on Days 1-7, and on Day 8 moxifloxacin 400 mg tablet and 2 macitentan-matching placebo tablets). Treatment B: macitentan 10 mg (1 macitentan 10 mg tablet and 2 placebo tablets once daily on Days 1-8). Treatment C: macitentan 30 mg (3 macitentan 10 mg tablets once daily on Days 1-8). Treatment D: placebo (3 placebo tablets on Days 1-8). There was a wash-out period of at least 10 days between the last study drug administration of the previous treatment and the first study drug administration of the following treatment.
  Interventions: Drug: Moxifloxacin 400 mg; Drug: Macitentan 10 mg; Drug: Macitentan 30 mg; Other: Placebo
- Treatment sequence ABDC (Experimental): Subjects received study medication in the sequence ABDC. Treatment A: moxifloxacin positive control (3 placebo tablets once daily on Days 1-7, and on Day 8 moxifloxacin 400 mg tablet and 2 macitentan-matching placebo tablets). Treatment B: macitentan 10 mg (1 macitentan 10 mg tablet and 2 placebo tablets once daily on Days 1-8). Treatment C: macitentan 30 mg (3 macitentan 10 mg tablets once daily on Days 1-8). Treatment D: placebo (3 placebo tablets on Days 1-8). There was a wash-out period of at least 10 days between the last study drug administration of the previous treatment and the first study drug administration of the following treatment.
  Interventions: Drug: Moxifloxacin 400 mg; Drug: Macitentan 10 mg; Drug: Macitentan 30 mg; Other: Placebo
- Treatment sequence DACB (Experimental): Subjects received study medication in the sequence DACB. Treatment A: moxifloxacin positive control (3 placebo tablets once daily on Days 1-7, and on Day 8 moxifloxacin 400 mg tablet and 2 macitentan-matching placebo tablets). Treatment B: macitentan 10 mg (1 macitentan 10 mg tablet and 2 placebo tablets once daily on Days 1-8). Treatment C: macitentan 30 mg (3 macitentan 10 mg tablets once daily on Days 1-8). Treatment D: placebo (3 placebo tablets on Days 1-8). There was a wash-out period of at least 10 days between the last study drug administration of the previous treatment and the first study drug administration of the following treatment.
  Interventions: Drug: Moxifloxacin 400 mg; Drug: Macitentan 10 mg; Drug: Macitentan 30 mg; Other: Placebo
- Treatment sequence CDBA (Experimental): Subjects received study medication in the sequence CDBA. Treatment A: moxifloxacin positive control (3 placebo tablets once daily on Days 1-7, and on Day 8 moxifloxacin 400 mg tablet and 2 macitentan-matching placebo tablets). Treatment B: macitentan 10 mg (1 macitentan 10 mg tablet and 2 placebo tablets once daily on Days 1-8). Treatment C: macitentan 30 mg (3 macitentan 10 mg tablets once daily on Days 1-8). Treatment D: placebo (3 placebo tablets on Days 1-8). There was a wash-out period of at least 10 days between the last study drug administration of the previous treatment and the first study drug administration of the following treatment.
  Interventions: Drug: Moxifloxacin 400 mg; Drug: Macitentan 10 mg; Drug: Macitentan 30 mg; Other: Placebo
- Treatment sequence DBAC (Experimental): Subjects received study medication in the sequence DBAC. Treatment A: moxifloxacin positive control (3 placebo tablets once daily on Days 1-7, and on Day 8 moxifloxacin 400 mg tablet and 2 macitentan-matching placebo tablets). Treatment B: macitentan 10 mg (1 macitentan 10 mg tablet and 2 placebo tablets once daily on Days 1-8). Treatment C: macitentan 30 mg (3 macitentan 10 mg tablets once daily on Days 1-8). Treatment D: placebo (3 placebo tablets on Days 1-8). There was a wash-out period of at least 10 days between the last study drug administration of the previous treatment and the first study drug administration of the following treatment.
  Interventions: Drug: Moxifloxacin 400 mg; Drug: Macitentan 10 mg; Drug: Macitentan 30 mg; Other: Placebo
- Treatment sequence ADCB (Experimental): Subjects received study medication in the sequence ADCB. Treatment A: moxifloxacin positive control (3 placebo tablets once daily on Days 1-7, and on Day 8 moxifloxacin 400 mg tablet and 2 macitentan-matching placebo tablets). Treatment B: macitentan 10 mg (1 macitentan 10 mg tablet and 2 placebo tablets once daily on Days 1-8). Treatment C: macitentan 30 mg (3 macitentan 10 mg tablets once daily on Days 1-8). Treatment D: placebo (3 placebo tablets on Days 1-8). There was a wash-out period of at least 10 days between the last study drug administration of the previous treatment and the first study drug administration of the following treatment.
  Interventions: Drug: Moxifloxacin 400 mg; Drug: Macitentan 10 mg; Drug: Macitentan 30 mg; Other: Placebo
- Treatment sequence CABD (Experimental): Subjects received study medication in the sequence CABD . Treatment A: moxifloxacin positive control (3 placebo tablets once daily on Days 1-7, and on Day 8 moxifloxacin 400 mg tablet and 2 macitentan-matching placebo tablets). Treatment B: macitentan 10 mg (1 macitentan 10 mg tablet and 2 placebo tablets once daily on Days 1-8). Treatment C: macitentan 30 mg (3 macitentan 10 mg tablets once daily on Days 1-8). Treatment D: placebo (3 placebo tablets on Days 1-8). There was a wash-out period of at least 10 days between the last study drug administration of the previous treatment and the first study drug administration of the following treatment.
  Interventions: Drug: Moxifloxacin 400 mg; Drug: Macitentan 10 mg; Drug: Macitentan 30 mg; Other: Placebo
- Treatment sequence BCDA (Experimental): Subjects received study medication in the sequence BCDA. Treatment A: moxifloxacin positive control (3 placebo tablets once daily on Days 1-7, and on Day 8 moxifloxacin 400 mg tablet and 2 macitentan-matching placebo tablets). Treatment B: macitentan 10 mg (1 macitentan 10 mg tablet and 2 placebo tablets once daily on Days 1-8). Treatment C: macitentan 30 mg (3 macitentan 10 mg tablets once daily on Days 1-8). Treatment D: placebo (3 placebo tablets on Days 1-8). There was a wash-out period of at least 10 days between the last study drug administration of the previous treatment and the first study drug administration of the following treatment.
  Interventions: Drug: Moxifloxacin 400 mg; Drug: Macitentan 10 mg; Drug: Macitentan 30 mg; Other: Placebo

INTERVENTIONS:
Drug: Moxifloxacin 400 mg
Drug: Macitentan 10 mg
  Other Names: Opsumit
Drug: Macitentan 30 mg
  Other Names: Opsumit
Other: Placebo

SUMMARY:
The study is intended to demonstrate that macitentan does not have an effect on cardiac repolarization exceeding the threshold of regulatory concern after repeated administration of daily oral doses of 10 and 30 mg to healthy male and female subjects.

ELIGIBILITY:
Inclusion Criteria:

* Ability to communicate well with the investigator in the local language, and to understand and comply with the requirements of the study.
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice and the local legislation.
* Males and females aged ≥ 18 and ≤ 55 years at screening.
* Women of childbearing potential must have had a negative pre-treatment serum pregnancy test and used consistently and correctly 2 methods of contraception at the same time from screening and up to 30 days after study treatment discontinuation. Abstinence was not considered a reliable method of contraception.
* Healthy on the basis of medical history and the assessments performed at screening.
* Physical examination without clinically relevant abnormalities at screening.
* Body mass index (BMI) ≥ 18.0 and ≤ 28.0 kg/m^2 at screening. Body weight at least 50.0 kg.
* Negative results from urine drug screen and alcohol test at screening.
* Willing and able to refrain from alcohol consumption from study start to the end of the study.
* Negative human immunodeficiency virus (HIV) serology and hepatitis serology at screening.
* Systolic blood pressure (SBP) 100-145 mmHg, diastolic blood pressure (DBP) 50-90 mmHg, and heart rate (HR) 45-90 bpm (all inclusive), measured on the dominant arm (dominant arm = writing arm).
* 12-lead ECG without clinically relevant abnormalities at screening and on Day 1 prior to drug administration.
* Hematology, blood chemistry, and urinalysis results not deviating from the normal range to a clinically relevant extent at screening and on Day 1 prior to drug administration.

Exclusion Criteria:

* Known hypersensitivity to any excipients of the drug formulations.
* Treatment with macitentan or another investigational drug in the 3 months prior to screening.
* History or clinical evidence of any disease and/or the existence of any surgical or medical condition, which might have interfered with the absorption, distribution, metabolism, or excretion of macitentan and moxifloxacin (except appendectomy and herniotomy).
* History or clinical evidence of drug abuse, alcoholism, or psychiatric disease within the 3 year period prior to screening.
* Caffeine consumption ≥ 800 mg per day at screening.
* History of fainting, collapse, syncope, blackouts, orthostatic hypotension, or vasovagal reactions.
* Chronic or relevant acute infections.
* History of relevant allergy/hypersensitivity.
* Previous treatment with any prescribed or over-the-counter medications or herbal remedies (including herbal medicines such as St John's Wort) within 2 weeks prior to first dosing or during the trial.
* Smoking and use of tobacco substitutes or nicotine substitutes.
* Loss of 250 mL or more blood in the 3 months prior to dosing (including blood donation).
* Positive results from the hepatitis serology at screening, except for vaccinated subjects.
* Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) above the upper limit of normal prior to randomization.
* Excessive physical activities within 1 week prior to randomization.
* Any cardiac condition (including ECG abnormalities) or illness with a potential to increase the cardiac risk of the subject or that might affect the corrected QT analysis (QTc).
* QTc > 450 ms or > 470 ms (using the ECG machine heart rate-correction method) before randomization for male or female subjects, respectively.
* Subjects with personal or family history of long-QT syndrome or hypokalemia.
* Legal incapacity or limited legal capacity at screening.
* Veins unsuitable for intravenous (i.v.) puncture on either arm (e.g., veins that are difficult to locate, access or puncture; veins with a tendency to rupture during or after puncture).
* Vulnerable subjects (e.g., persons kept in detention).
* Employee of the investigator or study center, with direct involvement in the proposed study or other studies under the direction of that investigator or study center, as well as family members of the employees or the investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2011-08; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Baseline-adjusted placebo-corrected QT interval according to Fridericia's correction (QTcF) | Day 8
  The QTcF interval was obtained directly from the Holter ECG monitoring.Triplicate ECG recordings were obtained from a 12-lead Holter recording device at various time points on Day 8. Baseline data were obtained from the pre-dose recording on Day 1 (from about 45 to 15 minutes prior to the morning dose). The QTcF interval is the QT interval (interval from beginning of the Q wave until end of the T wave) corrected for heart rate with Fridericia's formula (QTcF = QT/RR^0.33 where RR is 60/heart rate)

SECONDARY OUTCOMES:
Placebo corrected change from baseline in heart rate on Day 8 | Day 8
  Heart rate was obtained directly from the Holter ECG monitoring. Triplicate ECG recordings were obtained from a 12-lead Holter recording device at various time points on Day 8. Baseline data were obtained from the pre-dose recording on Day 1 (from about 45 to 15 minutes prior to the morning dose).
Placebo corrected change from baseline in RR interval (the interval from the onset of one QRS complex to the onset of the next QRS complex) on Day 8 | Day 8
  The RR interval was obtained directly from the Holter ECG monitoring. Triplicate ECG recordings were obtained from a 12-lead Holter recording device at various time points on Day 8. Baseline data were obtained from the pre-dose recording on Day 1 (from about 45 to 15 minutes prior to the morning dose).
Placebo corrected change from baseline in PR interval (time interval from the beginning of the P wave to the beginning of the QRS complex) on Day 8 | Day 8
  The PR interval was obtained directly from the Holter ECG monitoring. Triplicate ECG recordings were obtained from a 12-lead Holter recording device at various time points on Day 8. Baseline data were obtained from the pre-dose recording on Day 1 (from about 45 to 15 minutes prior to the morning dose).
Placebo corrected change from baseline in QRS interval (time interval from the beginning of the Q wave to the end of the S wave) on Day 8 | Day 8
  The QRS interval was obtained directly from the Holter ECG monitoring. Triplicate ECG recordings were obtained from a 12-lead Holter recording device at various time points on Day 8. Baseline data were obtained from the pre-dose recording on Day 1 (from about 45 to 15 minutes prior to the morning dose).
Number of participants with treatment emergent ECG abnormalities | 8 Days
  ECG were obtained from continuous 12-lead Holter ECG recordings. Morphological analyses were performed with regard to the ECG waveform interpretation for the following abnormalities: second degree heart block, third degree heart block, complete right bundle branch block, complete left bundle branch block, ST-segment change (elevation and depression separately), T-wave abnormalities (negative T waves only), and myocardial infarction pattern, and any new abnormal U waves.
Maximum plasma concentration (Cmax) of macitentan on Day 8 | Day 8
  Blood samples for pharmacokinetic analysis taken immediately prior to dosing with macitentan, and at 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 16, and 24 hours after dosing. Cmax was calculated on the basis of the blood sampling time points.
Maximum plasma concentration (Cmax) of the macitentan metabolite ACT-132577 on Day 8 | Day 8
  Blood samples for pharmacokinetic analysis taken immediately prior to dosing with macitentan, and at 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 16, and 24 hours after dosing. Cmax was calculated on the basis of the blood sampling time points.
Time to reach maximum plasma concentration (tmax) of macitentan on Day 8 | Day 8
  Blood samples for pharmacokinetic analysis taken immediately prior to dosing with macitentan, and at 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 16, and 24 hours after dosing. tmax was calculated on the basis of the blood sampling time points.
Time to reach maximum plasma concentration (tmax) of the macitentan metabolite ACT-132577 on Day 8 | Day 8
  Blood samples for pharmacokinetic analysis taken immediately prior to dosing with macitentan, and at 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 16, and 24 hours after dosing. tmax was calculated on the basis of the blood sampling time points.
Area under the plasma concentration-time curve over a dosing interval (AUCτ) of macitentan on Day 8 | Day 8
  Blood samples for pharmacokinetic analysis taken immediately prior to dosing with macitentan, and at 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 16, and 24 hours after dosing. AUCτ was calculated using the linear trapezoidal rule using the measured concentration-time values above the limit of quantification from time 0 to 24 hours after drug administration.
Area under the plasma concentration-time curve over a dosing interval (AUCτ) of the macitentan metabolite ACT-132577 on Day 8 | Day 8
  Blood samples for pharmacokinetic analysis taken immediately prior to dosing with macitentan, and at 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 16, and 24 hours after dosing. AUCτ was calculated using the linear trapezoidal rule using the measured concentration-time values above the limit of quantification from time 0 to 24 hours after drug administration.
Change from baseline to Day 8 in systolic blood pressure (SBP) | 8 days
  SBP was measured using an automatic oscillometric device, always on the dominant arm (i.e., dominant arm right = writing with right hand). Measurements were taken from the subject in a supine position after having rested for a 10-minute period.
Change from baseline to Day 8 in diastolic blood pressure (DBP) | 8 days
  DBP was measured using an automatic oscillometric device, always on the dominant arm (i.e., dominant arm right = writing with right hand). Measurements were taken from the subject in a supine position after having rested for a 10-minute period.
Change from baseline to Day 8 in heart rate | 8 days
  Heart rate was measured using an automatic oscillometric device, always on the dominant arm (i.e., dominant arm right = writing with right hand). Measurements were taken from the subject in a supine position after having rested for a 10-minute period.
Change from baseline to Day 8 in body weight | 8 days
  Body weight was measured using the same weighing scale for all subjects and throughout the study. The weighing scale had a precision of at least 0.5 kg.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Lindegger, PhD, Study Director — Actelion